CLINICAL TRIAL: NCT06627478
Title: Single-dose, Double-blind, Randomized, Three-period, Three-treatment, Six-sequence, Crossover Study to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity Between NKF-INS(G), US-Lantus®, and EU-Lantus®
Brief Title: Study to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity Between NKF-INS Glargine (G), United States (US)-Lantus®, and European Union (EU)-Lantus®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NKF-INS(G)-101
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- United States (US)-Lantus® (Active Comparator): Single subcutaneous dose administered over three treatment periods
  Interventions: Drug: US-Lantus®
- European Union (EU)-Lantus® (Active Comparator): Single subcutaneous dose administered over three treatment periods
  Interventions: Drug: EU-Lantus®
- NKF-INS Glargine (G) (Experimental): Single subcutaneous dose administered over three treatment periods
  Interventions: Drug: NKF-INS(G)

INTERVENTIONS:
Drug: NKF-INS(G) — Single subcutaneous dose of 0.5 IU/kg administered over three periods
  Arms: NKF-INS Glargine (G)
Drug: US-Lantus® — Single subcutaneous dose of 0.5 IU/kg administered over three periods
  Arms: United States (US)-Lantus®
Drug: EU-Lantus® — Single subcutaneous dose of 0.5 IU/kg administered over three periods
  Arms: European Union (EU)-Lantus®

SUMMARY:
Single-dose, double-blind, randomized, three-period, three-treatment, six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS Glargine (G), United States (US)-Lantus®, and European Union (EU)-Lantus®

DETAILED DESCRIPTION:
A single center, single-dose, double-blind, randomized, three-period, three-treatment, six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS(G), US-Lantus®, and EU-Lantus® using the euglycemic clamp technique in healthy male adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the participant.
2. Healthy male participants
3. Age between 18 and 50 years, both inclusive
4. Body Mass Index between 18.5 and 29.0 kg/m2, both inclusive
5. Body weight ≥ 59 kg
6. Fasting glucose concentration ≤ 5.5 mmol/L at screening
7. Considered generally healthy upon completion of medical history, physical examination, vital signs, electrocardiogram (ECG), and analysis of laboratory safety variables, as judged by the Investigator
8. Willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
9. Participants must agree to use condoms during sexual intercourse. Additionally, female partners of male participants should use highly effective contraception. All contraceptive measures apply from screening until 90 days after study treatment. Male participants must refrain from donating or banking sperm for 90 days after administration of study treatment.
10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

Exclusion Criteria:

1. Positive for human insulin antibodies at Screening
2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.
3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin, or any specific investigational product safety concern.
4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.
5. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.
6. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
7. Clinically significant abnormal ECG at screening.
8. Glycemia level ≥140 mg/dL 2 hours after the glucose load.
9. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
10. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.
11. Show evidence of an acute infection with fever or infectious disease at the time of enrollment.
12. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening.
13. Have positive test results for hepatitis B surface antigen (HBsAg), immunoglobulin M (IgM) antibody to hepatitis B core antigen (anti-HBc), or hepatitis C virus (HCV) antibodies at screening.
14. Intend to use over-the-counter medication within 7 days or prescription medication within 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement).
15. Have donated blood or had a blood loss of 500 mL 3 months prior to study enrollment.
16. Have an average weekly alcohol intake that exceeds 21 units per week or is unwilling to stop alcohol consumption from 48 hours prior to each dosing until being discharged from the Clinical Research Unit (CRU).
17. Employees or close relatives of the Sponsor, contract research organization (CRO), third-party vendors. or affiliates of the above-mentioned parties.
18. Inadequate venous access.
19. Vulnerable populations, e.g., persons in detention.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
To compare the Pharmacokinetic (PK) of NKF-INS Glargine(G) to United States (US)-approved and European Union (EU)-authorized Lantus to demonstrate PK similarity for metabolite 21A-Gly-human insulin (M1) | 60 and 0 minutes pre-dose and 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours post-dose
  Area Under the Curve (AUC)0-24h of M1

SECONDARY OUTCOMES:
To evaluate additional PK parameters of NKF-INS(G), US-approved and EU-authorized Lantus to demonstrate similarity for insulin glargine | 60 and 0 minutes pre-dose and 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours post-dose
  PK parameters for plasma insulin glargine concentrations and/or M1: maximum observed plasma exogenous insulin glargine concentration.
To evaluate additional PK parameters of NKF-INS(G), US-approved and EU-authorized Lantus to demonstrate similarity for M1 | 60 and 0 minutes pre-dose and 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours post-dose
  M1: maximum observed plasma exogenous insulin glargine concentration (Cmax), AUC0-24h, AUC0-6h, AUC6-12h, AUC0-12h, AUC12-18h, AUC18-24h, and AUC12-24h (fractional area under the plasma concentration-time curve), time to maximum plasma exogenous insulin glargine concentration (Tmax), AUC0-∞
To compare the Pharmacodynamic (PD) of NKF-INS(G) to US-approved and EU-authorized Lantus by examining glucose infusion rate (GIR) profiles after a single subcutaneous (SC) dose. | Time Frame: 60 and 0 minutes pre-dose and 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours post-dose
  GIRAUC0-24h, GIRAUC0-end of clamp, GIRAUC0-∞, GIRAUC0-6h, GIRAUC6-12h, GIRAUC0-12h, GIRAUC12-18h, GIRAUC18-24h, and GIRAUC12-24h (fractional area under the GIR-time curve), GIRmax, Total(T)GIRmax, and total amount of glucose infused during clamp procedure (Gtot)
To assess the safety of NKF-INS(G) | Day 1 to 7 weeks
  Adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- FARMOVS Clinical Research Organisation, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: No